CLINICAL TRIAL: NCT04239859
Title: Outcomes With Treatment and Withdraw of Secukinumab in Patients With Plaque Psoriasis Compared to Standard Care --- a Pragmatic Observational Study
Brief Title: Outcomes With Treatment and Withdraw of Secukinumab in Patients With Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Translational Immunology Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PsO1
Record Dates: First submitted 2019-12-04; First posted 2020-01-27 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — secukinumab; Methotrexate; Cyclosporine; Acitretin

STUDY DESIGN:
Intervention Model Description: To evaluate the real-life effectiveness of secukinumab as first-line systemic treatment in participants with moderate to severe PsO, the investigators would recruit a pragmatic control arm.
  ⦁ Intervention arm Eligible participants will be offered secukinumab as first-line systemic treatment for PsO. Standard dose of subcutaneous secukinumab for moderate to severe PsO will be given at 300 mg at weeks 0, 1, 2, 3, and 4, then monthly thereafter, for a total duration of 6 months.
  Secukinumab will be withdrawn after 6 months. For some participants, there may be relapse of PsO. Relapses will be managed as per standard care.
  ⦁ Pragmatic control arm
  Eligible participants will be recruited to pragmatic control arm in these circumstances:
  * Patient disagree to secukinumab for personal reasons.
  * The quota for secukinumab is exhausted.
  * The management of PsO in this pragmatic control arm will be the same as that in the standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Secukinumab (Experimental): Participants will be offered secukinumab as first-line systemic treatment for moderate to severe PsO. The indication for secukinumab will be equivalent to current registered indications. Standard dose of subcutaneous secukinumab for moderate to severe PsO will be given at 300 mg at weeks 0, 1, 2, 3, and 4, then monthly thereafter, for a total duration of 6 months.
  secukinumab will be withdrawn after 6 months. For some participants, there may be relapse of PsO. Relapses will be managed as per standard care.
  Interventions: Biological: secukinumab
- Standard Care (Active Comparator): The management of PsO in the control arm will be the same as that in the standard care.
  The standard care for moderate to severe PsO in Singapore is to start either phototherapy, methotrexate, acitretin or cyclosporin A.
  Interventions: Drug: Methotrexate; Drug: Cyclosporin A; Drug: Acitretin

INTERVENTIONS:
Biological: secukinumab — Secukinumab for 6 months, given at weeks 0, 1, 2, 3 and 4, then monthly till 6 months. 300mg per administration, subcutaneously.
  Arms: Secukinumab
Drug: Methotrexate — Oral tablet up to 15mg per week
  Arms: Standard Care
Drug: Cyclosporin A — Oral capsule up to 200mg per day
  Arms: Standard Care
Drug: Acitretin — Oral capsule up to 25mg per day
  Arms: Standard Care

SUMMARY:
Psoriasis (PsO) is a systemic immune disease that affect 2-4% of the population worldwide. PsO causes tremendous burden in terms of quality of life, psychological impact, disability and work productivity of affected individuals. PsO is associated with an increased risk of cardiovascular morbidities and mortality in the long term. Up to 30% of PsO patients develop psoriatic arthritis (PsA) over time causing joint deformities and further disabilities. Majority of patients with PsA developed PsO first, and arthritis develop 5-10 years after. PsA and PsO are increasingly recognized as two entities under the umbrella of psoriatic diseases.

Advances in biological treatments have greatly improved the prognosis of patients with PsO. Remarkable efficacies have been demonstrated for patients with moderate to severe PsO in randomized controlled trials (RCTs). However, the high cost of biological treatment is one of the major barriers to its prescription and many patients may have limited access to these treatments.

The best treatment strategy for PsO that takes into account efficacy and cost effectiveness is unknown. For instance, whether some PsO patients can stop biological treatment and be treated with non-biologic medications upon relapse, which may enhance cost effectiveness of treatment. Preliminary studies have shown that some PsO patients were able to maintain good control of disease without medications after biologics withdrawal. The patho-immunological mechanisms behind long term remission after drug withdrawal is poorly understood. Better understanding of these mechanisms in maintaining remission and relapses will advance the development of biomarkers that eventually guide development of best treatment strategies for PsO.

Secukinumab targets interleukin (IL)-17a and is highly efficacious in the treatment of plague PsO with a favorable safety profile. Some patients may have the response maintained after withdrawal of secukinumab. With the proven efficacies, sustainability after withdrawal and safety profile, secukinumab could be a choice of initial treatment for patients with moderate to severe PsO. Secukinumab has been recommended as first line treatment for selected patients with moderate to severe PsO by the American Academy of Dermatology and the European S3 guidelines. However, the use of biologics as first line is limited by cost issue. Overall, real-life data on biologic treatment for moderate to severe PsO is scanty.

DETAILED DESCRIPTION:
First, the investigators hypothesize that a proportion of participants with moderate to severe PsO may sustain good outcomes when a short course of secukinumab is withdrawn.

Second, the investigators hypothesize that they can identify the perturbations in the architecture of the immunome which are pathogenic, and to discriminate such perturbations based on treatment and clinical responses, thus distilling therapeutics and diagnostics signatures.

Therefore, the objectives of this study are as follow:

Specific aim 1: To describe the clinical course, sustained good outcomes, relapse rate, time to relapse and quality of life in PsO participants who stopped a 6-month short course treatment of secukinumab, till the end of 2-years.

Specific aim 2: To identify the genomic and immunomics signatures in skin biopsies and blood in PsO participants who has good outcomes (PASI 75) at 6 months, comparing treatment vs pragmatic control.

Specific aim 3: To identify the genomic and immunomics signatures in skin biopsies and blood in PsO participants who sustained good outcomes at 1 year after stopping secukinumab, compared to those relapsed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>21-year-old).
* Diagnosed by dermatologist as plague-type PsO.
* Having moderate to severe plague-type PsO as defined by the following:
* Psoriasis Area and Severity Index (PASI) ≥12/72,
* And, investigator Global Assessment Score (IGA) ≥3,
* And, PsO involving body surface area involvement (BSA) ≥10%
* And Candidate for phototherapy and/or systemic therapy
* Topical corticosteroid up to moderate potencies are allowed
* Able to provide informed consent.

Exclusion Criteria:

* Forms of PsO other than plaque-type.
* Evidence of skin conditions at the time of the screening visit (e.g. eczema) that would interfere with evaluation of the effect of the investigational product on PsO.
* Evidence of active tuberculosis or other active infections (like Hepatitis C/B), malignancy; active or known use of other immunosuppressive drugs (eg. AIDS, rheumatoid arthritis, organ rejection etc) at the screening visit.
* Previous exposure to any systemic immunosuppressants (eg. methotrexate) or phototherapy
* History or current signs of a severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances.
* Having current or history of malignancy, except non-melanoma skin cancer, within the previous 5 years that have been adequately treated.
* History of inflammatory bowel disease.
* Pregnancy or lactating mothers.
* As treatment regimen is different, participants with evidence of PsA will be excl

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of secukinumab treated PsO participants free of relapse after secukinumab withdrawal | 12 months from secukinumab withdrawal or 18 months from baseline
  The investigators will describe the proportion of secukinumab treated PsO participants free of relapse at 12 months after secukinumab withdrawal.

SECONDARY OUTCOMES:
Proportion of secukinumab treated PsO participants free of relapse after secukinumab withdrawal | 15, 18, and 24 months from secukinumab withdrawal or 21, 24, and 30 months from baseline
  The investigators will describe the proportion of secukinumab treated PsO participants free of relapse at 15, 18, and 24 months after secukinumab withdrawal.
Proportion of participants achieving PASI 50 | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. PASI 50 indicates a 50% improvement of PASI scores.
Proportion of participants achieving PASI 75 | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. PASI 75 indicates a 75% improvement of PASI scores.
Proportion of participants achieving PASI 90 | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. PASI 90 indicates a 90% improvement of PASI scores.
Proportion of participants achieving clearance | 3 months and 6 months
  Psoriasis is assessed by using the Psoriasis Area Severity Index (PASI) that measures the severity (intensity of redness, thickness and scaling is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4)) and percentage of affected area in four regions of the body (head and neck, upper limbs, trunk, lower limbs, expressed as nil (0), 1-9% (1), 10-29% (2), 30-49% (3), 50-69% (4), 70-89% (5) or 90-100% (6)). The score ranges from 0 (no psoriasis) to 72 (severe psoriasis). Percentage of improvement of PASI at 3 month and 6 month time points will be calculated from baseline. Clearance indicates a 100% improvement of PASI scores.
Quality of life 1 (EuroQoL-5D-5L) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both secukinumab treated and standard care) the investigators will describe the following:
  Every 3-6 monthly till end of 30 months, investigators will evaluate the change scores of Quality of Life (EQ5D-5L). It consists of the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions. Each dimension is measured on a scale of 1-5, with '1' indicating no problem, '2' indicating slight problems, '3' indicating moderate problems, '4' indicating severe problems, and '5' indicating unable to/extreme problems. The highest and the lowest scores for both EQ-5D-5L indices were 1.00 (best imaginable health) and -0.769 respectively; where negative values are valued as worse than dead.
  EQ VAS records the patient's self-rated health on a vertical visual analogue scale from 0-100 with '0' indicating worst health one can imagine and '100' indicating best health one can imagine.
Quality of life 2 (Dermatology Life Quality Index - DLQI) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both secukinumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the change scores of Dermatology Life Quality Index (DLQI) at various time points from baseline. DLQI is measured on a scale of 0-3 or not relevant, with '0' indicating not relevant or not at all, '1' indicating a little, '2' indicating a lot, '3' indicating very much. The final score ranges from 0 (minimal effect on quality of life) to 30 (maximum effect on quality of life).
Quality of life 3 (Hospital Anxiety and Depression Scale - HADS) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both secukinumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the change scores of Hospital Anxiety and Depression Scale (HADS) at various time points from baseline. HADS is a 14 item scale with 7 of the items related to anxiety and the other 7 related to depression. Each item on the questionnaire is scored from 0-3, resulting in anxiety and depression scores each of 0 (no anxiety/depression) to 21 (severe anxiety/depression).
Patient Global Assessment | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both secukinumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the change scores of Patient Global Assessment (0-10) at various time points from baseline, with higher scores meaning worse outcome.
Patient Acceptable Symptom State (PASS) | 3, 6, 9, 12, 15, 18, 24 and 30 months
  In all participants (both secukinumab treated and standard care) the investigators will describe the following:
  - Questionnaires on health status and quality of life every 3-6 monthly till end of 30 months.
  The investigators will evaluate the proportion of patient defined acceptable state (acceptable/unacceptable) and whether the symptoms are worse than usual (yes/no) at various time points from baseline.
Proportion of participants in secukinumab treatment arm maintaining PASI 50 after secukinumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the secukinumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI 50 at 3, 6, 12, 18 and 24 months after stopping secukinumab treatment
Proportion of participants in secukinumab treatment arm maintaining PASI 75 after secukinumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the secukinumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI 75 at 3, 6, 12, 18 and 24 months after stopping secukinumab treatment
Proportion of participants in secukinumab treatment arm maintaining PASI 90 after secukinumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the secukinumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI 90 at 3, 6, 12, 18 and 24 months after stopping secukinumab treatment
Proportion of participants in secukinumab treatment arm maintaining clearance after secukinumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the secukinumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants maintaining PASI clearance at 3, 6, 12, 18 and 24 months after stopping secukinumab treatment
Proportion of participants in secukinumab treatment arm flaring after secukinumab withdrawal | 9, 12, 18, 24 and 30 months from baseline
  For participants in the secukinumab treatment arm, the investigators describe the following in additional:
  - The proportion of participants who flare (defined as losing the PASI50 response) at 3, 6, 12, 18 and 24 months after stopping secukinumab treatment
Histological changes in the skin biopsies of participants in secukinumab treatment arm who relapsed after secukinumab withdrawal (or at 18 months if no relapse) | Baseline, 6 months, at relapse (or 18 months if no relapse)
  For participants in the secukinumab treatment arm, the investigators will evaluate the following outcomes at relapse (or at 12 months after stopping secukinumab if no relapse):
  - Histological sections of morphologically psoriasis (lesional) and morphologically no psoriasis (nonlesional) skin biopsies. Skin biopsies at relapse will be scored for the degree of histological improvement compared to that participant's disease at 6 months on a five point scale; -1 (worse) to +3 (excellent).
Skin genomic profiles in the skin biopsies of participants in secukinumab treatment arm who relapsed after secukinumab withdrawal (or at 18 months if no relapse) | Baseline, 6 months, at relapse (or 18 months if no relapse)
  For participants in the secukinumab treatment arm, the investigators will evaluate the following outcomes at relapse (or at 12 months after stopping secukinumab if no relapse):
  - Whole RNA genome transcriptome of the skin biopsies will be studied. The change in transcriptomes at relapse compared to 6-month will be evaluated.
Peripheral blood immunome profiles of participants in secukinumab treatment arm who relapsed after secukinumab withdrawal (or at 18 months if no relapse) | Baseline, 6 months, at relapse (or 18 months if no relapse)
  For participants in the secukinumab treatment arm, the investigators will evaluate the following outcomes at relapse (or at 12 months after stopping secukinumab if no relapse):
  * The B-cell and T-cell subtypes in the peripheral blood will be evaluated using mass cytometry, and compared to that of baseline and 6 months.
  * The investigators will evaluate the change in B-cell and T-cell Subtypes at relapse compared to baseline and 6 months.
Histological changes in the skin biopsies | Baseline and 6 months
  In all participants, the investigators will evaluate the skin genomic profiles that differentiate between secukinumab versus standard care control arms.
  - Histological sections of morphologically psoriasis (lesional) and morphologically no psoriasis (non lesional) skin biopsies at baseline and 6 months will be examined. Skin biopsies at 6 month will be scored for the degree of histological improvement compared to that participant's baseline disease on a five point scale; -1 (worse) to +3 (excellent).
Skin genomic profiles | Baseline and 6 months
  In all participants, the investigators will evaluate the skin genomic profiles that differentiate between secukinumab versus standard care control arms.
  - Whole RNA genome transcriptome of the skin biopsies will be studied. The change in transcriptomes at 6 months compared to baseline will be evaluated.
Peripheral blood immunome profiles | Baseline and 6 months
  In all participants, the investigators will evaluate the blood immunome profiles that differentiate between secukinumab versus standard care control arms.
  - The B-cell and T-cell subtypes in the peripheral blood of participants in both secukinumab and standard care arms will be evaluated using mass cytometry. - The investigators will evaluate the change in B-cell and T-cell subtypes at 6 months from baseline for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ying Leung, MD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Outram Park, Singapore

IPD SHARING:
Plan to Share IPD: No